CLINICAL TRIAL: NCT05308017
Title: Does Sheath Size Matter? Wolf 24 F vs. Storz 28 F Laser Sheath Size for Holmium Laser Enucleation of the Prostate
Brief Title: Wolf 24 F vs. Storz 28 F Laser Sheath Size for HoLEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Krambeck, Director of the Endourology/Stone Division, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00215646
Record Dates: First submitted 2022-03-06; First posted 2022-04-01 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Benign Prostatic Hypertrophy
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: randomized to one of two different types of scopes.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Richard Wolf 24F Laser scope (Active Comparator)
  Interventions: Device: Richard Wolf 24F Laser scope
- Karl Storz 28F Laser scope (Active Comparator)
  Interventions: Device: Karl Storz 28F Laser Scope

INTERVENTIONS:
Device: Richard Wolf 24F Laser scope — 24F Laser with HoLEP
  Arms: Richard Wolf 24F Laser scope
Device: Karl Storz 28F Laser Scope — 28 F Laser with HoLEP
  Arms: Karl Storz 28F Laser scope

SUMMARY:
The purpose of this study is to compare two different types of scopes that can be used for HoLEP. HoLEP is performed through the urethra using a Laser scope to remove obstructing prostate tissue. Laser scopes come in different sizes (diameters).

ELIGIBILITY:
Inclusion Criteria:

* Patients Males 18-89 undergoing HoLEP for the treatment of bothersome lower urinary tract symptoms

Exclusion Criteria:

* Patients who lack decisional capacity

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male only
Enrollment: 152 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Surgery Time difference between the 24F laser scope and the 28F laser scope | Day 0
  comparing operative time between the 24F and the 28F laser scope groups.

SECONDARY OUTCOMES:
Surgeon evaluation of Laser scopes flow rate | Day 0
  Internal survey within REDCap to be completed by the surgeon using the scope. The survey will ask the surgeon the following questions after every surgery
  1) How was the flow through the scope?
  a. 1) Poor 2) Problematic 3) Mediocre 4) Adequate 5) Good
Surgeon evaluation of Laser scope visualization | Day 0
  Internal survey within REDCap to be completed by the surgeon using the scope. The survey will ask the surgeon the following questions after every surgery
  2) How was the visualization?
  a. 1) Poor 2) Problematic 3) Mediocre 4) Adequate 5) Good
Surgeon evaluation of Laser scope bladder injury | Day 0
  Internal survey within REDCap to be completed by the surgeon using the scope. The survey will ask the surgeon the following questions after every surgery
  3) Did bladder injury occur?
  a. 1) Yes 2) No

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dean NS, Lee MS, Assmus MA, Guo J, Xu P, McDonald A, Fadl-Alla A, Helin J, Krambeck AE. Does Resectoscope Sheath Size Influence Holmium Laser Enucleation of the Prostate Outcomes? A Prospective Randomized Controlled Trial. J Endourol. 2023 Dec;37(12):1261-1269. doi: 10.1089/end.2023.0383. PMID 37786336